CLINICAL TRIAL: NCT03097510
Title: Meditation and Emotional Intelligence: A Randomized Controlled Trial
Brief Title: Meditation and Emotional Intelligence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: Center for Wellness and Achievement in Education (Unknown)
Responsible Party: Principal Investigator, Sanford Nidich, Associate Director, Maharishi University of Management Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLF-WEHF-1440
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Job Stress; Perceived Stress
Keywords: Perceived stress; Leadership; Transcendental Meditation
MeSH Terms: conditions — Occupational Stress | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: data collectors and investigators were blind to treatment status of the subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation (Experimental): The TM technique is a simple, natural, effortless technique that allows the mind to experience finer levels of the thinking process until the mind transcends and experiences the source of thought, a state of deep, integrated relaxation. During the meditation session, the active mind settles down to a silent yet fully awake state of awareness. TM was taught to study participants by certified instructors, using standardized procedures for teaching.
  Interventions: Behavioral: Transcendental meditation
- Wait list control (No Intervention): This wait list group served as the control group. After the study was completed, the wait-list controls were given the option to learn the TM technique as their reward for participating as controls during the 4 month study.

INTERVENTIONS:
Behavioral: Transcendental meditation — The TM technique was taught as a standard 7 step course over 4 consecutive days. Thereafter, subjects attended bimonthly group meetings for more advanced knowledge over the four month intervention period.
  Other Names: TM technique
  Arms: Transcendental Meditation

SUMMARY:
This randomized controlled trial evaluated the impact of the Transcendental Meditation program on emotional intelligence and perceived stress in supervisors and administrative staff in a public school system

DETAILED DESCRIPTION:
The objective of this study was to determine whether a mind-body technique, known as the practice of Transcendental Meditation® (TM), could significantly increase emotional intelligence and decrease perceived stress in supervisors and administrative staff in a public school system. For this purpose, 96 participants from the administrative offices of the San Francisco Unified School District were randomly assigned to either immediate start of the TM program or to a delayed start wait-list control group. Subjects learning TM were instructed to meditate for 20 minutes twice a day for the four month duration of the project. All subjects were administered the BarOn Emotional Quotient Inventory (EQ-i) and Perceived Stress Scale (PSS) at baseline and posttest. If successful, these findings would suggest that TM could be used as a professional development program in organizations to increase emotional intelligence and decrease perceived stress, in turn enhancing leadership capacity and organizational effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* an employee of the San Francisco Unified School District (SFUSD),
* attendance at an informational meeting on the TM program,
* willingness to be randomly assigned to either active treatment or the control group.

Exclusion Criteria:

* having already learned the TM program,
* not being available to attend treatment or testing sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Emotional Quotient Inventory (EQ-i) | Change from baseline EQ-i at four months
  The EQ-i is a self-report instrument that measures a range of non-cognitive capabilities, competencies, and skills that influence one's ability to succeed in coping with environmental demands and pressures.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Change from baseline PSS at four months
  The PSS is a 14-item instrument that measures the degree to which situations in one's life are appraised as stressful.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent D Valosek, Study Director — Center for Wellness and Achievement in Education

IPD SHARING:
Plan to Share IPD: Undecided
data may be available upon request from other researchers but at the discretion of the principal investigator